CLINICAL TRIAL: NCT01695343
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Repeat-dose Study of KB001-A in Subjects With Cystic Fibrosis Infected With Pseudomonas Aeruginosa
Brief Title: Study to Evaluate the Effect of KB001-A on Time-to-Need for Antibiotic Treatment
Acronym: KB001-A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Humanigen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KB001A-05
Record Dates: First submitted 2012-09-25; First posted 2012-09-27 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Pseudomonas aeruginosa (Pa); CF
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- KB001-A (Experimental): KB001-A administered up to 5x intravenously (IV) at 10 mg/kg up to a maximum dose of 800 mg per dose.
  Interventions: Biological: KB001-A
- Placebo Comparator (Placebo Comparator): Placebo administered up to 5x intravenously
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Biological: KB001-A
  Arms: KB001-A
Drug: Placebo Comparator
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to confirm and extend the Phase 1-2 KB001 findings of an airway anti-inflammatory effect in CF individuals with chronic Pseudomonas aeruginosa (Pa) airway infection. It is hypothesized that steady-state levels of KB001-A in CF subjects with airway Pa infection will be safe and well-tolerated, and will increase the time-to-need for antibiotic treatment (IV, inhaled, or oral) for worsening of respiratory tract signs and symptoms compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with CF who are older than 50 years of age may participate if treated with 2 or more courses of antibiotics (IV and/or oral) for respiratory sign and symptoms (CF exacerbation) in the 12 months before the Screening Visit
* Confirmed diagnosis of CF
* At least 2 respiratory tract cultures in the previous 12 months, with Pa present. The most recent positive Pa culture must be within 12 weeks before the Screening Visit (or obtain a positive culture at screening)
* FEV1 % levels within acceptable ranges (per the study protocol)
* Received inhaled ABX for equivalent of 8 weeks or greater in the 26 weeks before the Day 0 Visit

Exclusion Criteria:

* Treatment with antibiotics for acute illness within the 4 weeks before the Day 0 Visit
* Use of systemic corticosteroids within the 4 weeks before the Day 0 Visit
* Any change in regimen of CF maintenance therapies within the 4 weeks before the Day 0 Visit
* History of sputum cultures positive for B. cepacia complex in the 2 years before the Screening Visit
* History of organ transplantation
* Current smoker (tobacco, marijuana, or any other material). Use of smokeless inhalers/vaporizers for these materials is also prohibited
* History of drug addiction or alcohol abuse in the 12 months before the Screening Visit
* History of hepatic disease (clinical cirrhosis or portal hypertension), renal dysfunction
* Breast-feeding or pregnancy as evidenced by a positive blood pregnancy test
* Receiving any investigational drug in the 16 weeks (or 5 half lives) before the Day 0 Visit, whichever is longer

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 182 (Actual)
Dates: Start 2012-12; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of KB001-A on time-to-need for antibiotic (ABX) treatment for worsening of respiratory tract signs and symptoms. | 16 Weeks
  Time-to-need for ABX treatment will be the length of time between study material dosing and administration of ABX as needed for worsening respiratory conditions.

SECONDARY OUTCOMES:
Safety and tolerability of KB001-A | 16 Weeks
  Safety and tolerability will be measured by Adverse Events (AEs) and laboratory assessments

CONTACTS AND LOCATIONS:
Overall Officials: Nestor A. Molfino, MD., MSc, Study Chair — KaloBios Pharmaceuticals, Inc.
Locations (64):
- United States (55):
  - Mobile, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Long Beach, California
  - Oakland, California
  - Orange, California
  - Stanford, California
  - Aurora, Colorado
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Boise, Idaho
  - Glenview, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Portland, Maine
  - Boston, Massachusetts
  - Worchester, Massachusetts
  - Detriot, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Hanover, New Hampshire
  - Manchester, New Hampshire
  - Albuquerque, New Mexico
  - Albany, New York
  - Hawthorne, New York
  - New Hyde Park, New York
  - New York, New York
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Colchester, Vermont
  - Richmond, Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Australia (3):
  - New Lambton, New South Wales
  - Parkville, Victoria
  - Nedlands, Western Australia
- Israel (4):
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Tel Litwinsky
- New Zealand (2):
  - Dunedin
  - Hamilton